CLINICAL TRIAL: NCT02544386
Title: Impact of Hemiplegia Due to Stroke on the Microarchitecture of the Bone: Evaluation Using Micro CT 3D High Resolution and by Magnetic Resonance Imaging (MRI)
Brief Title: Impact of Hemiplegia Due to Stroke on the Microarchitecture of the Bone
Status: Terminated | Type: Observational
Why Stopped: Inclusion rhythm too slow
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 0701116; 2008-A00048-47 (Other: AFFSAPS)
Record Dates: First submitted 2015-09-07; First posted 2015-09-09 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Stroke; Hemiplegia
Keywords: bone microarchitecture; hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients who have experienced a vascular hemiplegia and accept bone measure by MRI and 3D CT scan
  Interventions: Procedure: MRI and 3D CT scan

INTERVENTIONS:
Procedure: MRI and 3D CT scan — Measurement of bone microarchitecture at the legs and wrists by 3D CT Scan and measuring the proportion of fat in the imaging leg bone (MRI)

SUMMARY:
In hemiplegic, there is very little data on the impact of neurological deficit on the microarchitecture independent of bone mineral density and composition of the bone marrow. Rare studies have shown the relationship between some micro-architectural parameters and severity of neurological deficit. There is no study in humans on the evolution of the parameters of the microarchitecture assessed by 3D micro-tomography in the early phase of the installation of neurological deficits after stroke, in terms of a bearing bone, tibia, that a non-load bearing bones, radius.

DETAILED DESCRIPTION:
Each patient must answer several questionnaires about their calcium intake and its ability to perform everyday tasks. They will also have 3 blood samples (15 ml each time), 3 measure of bone by 3D micro-tomography and 2 MRI examination. These examinations and sampling will take place after 30 days after stroke onset (except for MRI) and again after three months and six months after the stroke (the same day as the medical follow-up visit).

ELIGIBILITY:
Inclusion criteria

* at least 30 years
* vascular hemiplegia
* National Institute of Health Stroke Score equal 4 or greater with a motor of upper limb score greater than or equal 2 and a motor score of greater than or equal legs 2

Exclusion criteria

* Concomitant bone disease
* Endocrinopathies
* Phasic disorders understanding
* Contra-indication to MRI

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient aged at least 30 who have experienced a vascular hemiplegia within 30 days before enrollment
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Bone volume / tissue volume | 90 days
  Measure of Bone volume / tissue volume by the 3D CT scan

SECONDARY OUTCOMES:
Bone volume / tissue volume | 1 day
  Measure of Bone volume / tissue volume by the 3D CT scan
intraosseous fat | 90 days
  Measure the percentage of the intraosseous fat by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Thierry THOMAS, MD-PhD, Principal Investigator — CHU SAINT-ETIENNE